CLINICAL TRIAL: NCT05551962
Title: Comparative Analysis of the Effectiveness of Various Methods of Increasing the Thickness of Soft Tissues During Dental Implantation in the Esthetic Zone of the Maxilla
Brief Title: Increasing the Thickness of Soft Tissues in the Esthetic Zone Around Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10012022
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Soft Tissue Atrophy
Keywords: connective tissue graft; xenogeic collagen matrix; increasing of soft tissue thickness; dental implant; soft tissue augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First group (Active Comparator): The patients undergo implant placement in combination with an increase in the thickness of soft tissues using a free connective tissue graft from the tuber region on the maxilla or palate.
  Interventions: Procedure: Soft tissue augmentation with CTG
- Second group (Experimental): The patients undergo implant placement in combination with an increase in the thickness of soft tissues using collagen matrix "Fibro-Gide"
  Interventions: Procedure: Soft tissue augmentation with CM

INTERVENTIONS:
Procedure: Soft tissue augmentation with CTG — 1. Incision the mucosa at the alveolar ridge, mucosal-periosteal flap elevation
  2. Placement of the Astra Tech dental implant (Dentsply, Germany)
  3. Sampling of free connective tissue graft from the maxilla tuber area
  4. Fixation of the graft to the vestibular flap
  5. Suturing the wound tightly
  Arms: First group
Procedure: Soft tissue augmentation with CM — 1. Incision the mucosa at the alveolar ridge, mucosal-periosteal flap elevation
  2. Placement of the Astra Tech dental implant (Dentsply, Germany)
  3. Modeling of sterile collagen matrix according to the shape of the recipient bed
  4. Fixation of the collagen matrix to the vestibular flap
  5. Suturing the wound tightly
  Arms: Second group

SUMMARY:
This is an interventional prospective randomized clinical trial (RCT) in parallel groups. This study is aimed at detecting a difference in the increase in the thickness of soft tissues of at least 0.3 mm between the two groups (the standard deviation [SD] of 0.3 mm and the average value of 1.2 mm was borrowed from an article published by Cairo F et al., 2017). Using SampleSizeCalculator, it was calculated that the number of patients in each group should be 14 (alpha = 0.05; power = 80%). This number was increased by 10%, taking into account possible exceptions from the study. The sample size is 30 patients who will be randomly divided into two groups depending on the surgical intervention used. First group - patients will undergo increasing the thickness of the mucous membrane using free connective tissue graft from tuberosity area of the maxilla or palate. Second group - patients will undergo increasing the thickness of the mucous membrane using collagen matrix "Fibro-Gide" (Geistlich Pharma AG, Bahnhofstrasse 40, 6110 Wolhusen, Switzerland; registration in Russia 19.08.2020 No FSZ-20207/11765). In the postoperative period the value of soft tissue thickness gain, severity of pain syndrome, collateral edema, Doppler flowmetry, probing depth, soft tissue aesthetics, keratinized mucosa width and quality of life will be assessed. In addition, after 3 months simultaneously with installation of gingiva formers biopsy specimens will be sampled with mucotome in the area of the intervention followed by histomorphometric analysis of the obtained biopsies.

DETAILED DESCRIPTION:
The aim of this research is to perform a comparative clinical and histomorphometric analysis of soft tissues in the area of soft tissue graft and collagen matrix transplantation. Thirty patients diagnosed with partial absence of teeth will be examined on the basis of the Department of Surgical Dentistry of the E.V. Borovsky Institute of Dentistry of I.M. Sechenov First Moscow State Medical University. Patients have a soft tissue thickness deficiency from the vestibular surface in the area of the planned dental implant placement in the esthetic zone of the maxilla, which is an indication for its increase. All patients will be randomly divided into two groups depending on method of soft tissue augmentation used. In 1 group (n=15) transplantation of a free connective tissue graft (CTG) from tuberosity area of the maxilla or palate is performed. In 2 group (n=15) collagen matrix "Fibro-Gide" will be used. According to gender and age characteristics, both groups will be comparable. Randomization of patients will be carried out at the stage of surgical intervention as follows: after a dental implant placement and preparation of recipient's bed, an envelope with a randomly assigned treatment method (using a connective tissue graft or a collagen matrix) will be opened.

During the operation, incision will be made along the top of the alveolar ridge within the defect; a full-thickness muco-periosteal flap will be elevated. Traditional 2-stage dental implantation is performed according to surgical protocols of dental implant systems Astra Tech (Dentsply Implants Manufacturing GmbH, Germany; registration in Russia 27.12.2019 No FSZ 2015/3214). A free connective tissue graft will be harvested in patients of the first group. Graft will be fixed with a horizontal U-shaped suture to the buccal muco-periosteal flap. In second patients group a fragment of the collagen matrix "Fibro-Gide" will be fixed to the buccal muco-periosteal flap (Geistlich Pharma AG, Bahnhofstrasse 40, 6110 Wolhusen, Switzerland; registration in Russia 19.08.2020 No FSZ - 20207/11765). For patients of all groups mobilization of the muco-periosteal flap conducts followed by suturing the wound tightly without tension with simple interrupted sutures.

Postoperative recommendations will include rinsing with 0.2% chlorhexidine gluconate mouthwash solution (Corsodyl, GlaxoSmithKline 77.99.11.915.Д.005285.07.03) twice a day for a week and receiving antibiotic (Amoxicillin + Clavulanic Acid, 1 g Amoxiclav, LEK, d.d., Slovenia, 22.07.2011, П N012124/01) twice a day for 5 days. To relieve pain, 100 mg of Nimesulide (Nise; Dr. Reddy's Laboratories Ltd., India, 26.05.2009, П N012824/03) will be prescribed. The stage of the implant uncovering with hilling abutments installation is carried out 3 months after the intervention. At this stage, a soft tissue fragment will be taken using a mucotome in the area of the previously performed mucous membrane thickness increasing for subsequent histomorphometric analysis. In the study we will use both conventional light microscopy (microscopy in the light field) and polarizing microscopy - to estimate the content of collagen fibers in preparations stained with picrosirius red. During a morphometric study we will carry out a quantitative assessment of the characteristics of the epithelial layer, the basement membrane relative length (the ratio of the absolute length of the basement membrane to the length of the epithelial layer), the characteristics of the underlying connective tissue.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of written informed consent of the patient to participate in the study;
2. Age from 18 to 45 years;
3. The presence of an included defect in the esthetic zone part of maxilla with a sufficient volume of bone tissue;
4. Soft tissue thickness <3 mm on the vestibular side;
5. Adjacent teeth without periodontal pathology, the depth of probing should not exceed 3 mm along the entire dentoalveolar furrow;
6. Satisfactory level of oral hygiene;
7. Patients without concomitant pathology or with concomitant pathology in the compensation stage.

Non-inclusion criteria:

1. Age less than 18 and more than 45 years;
2. Heavy smokers (more than 10 cigarettes a day);
3. Patients with somatic diseases in the stage of decompensation or in the stage of exacerbation;
4. Patients with malignant tumors, as well as patients with a history of radiation and chemotherapy over the past 5 years;
5. Taking medications that affect the healing of soft tissues (nonsteroidal anti-inflammatory drugs, steroid drugs);
6. Pregnancy and breastfeeding;
7. Patients with mental disorders.

Exclusion Criteria:

1. Patients with infections either periodontally or periapically, which developed after inclusion in the study;
2. Pregnancy following entrance into the study;
3. Patients having poor oral hygiene or not wanting to carry out oral hygiene measures;
4. Patients who, for one reason or another, could not complete the entire protocol to the end.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
The amount of soft tissue thickness gain | Day 90 compared to the 0th day (initial value)
  The value of the increase in the thickness of soft tissues in the study area (mm) on the 90th day compared to the 0th day (initial value).To carry out the measurement an optical impression will be taken using the Primescan intraoral scanner (Dentsply/SIRONA,Germany, 16.05.2019, № РД-27221/26851) before the operation and on the 90th day after the operation. Further, in the specialized program GOM Inspect the stl-files will be compared and the vestibular contour changes will be evaluated at 3 equidistant points in the coronary-apical direction.

SECONDARY OUTCOMES:
Assessment of the severity of pain syndrome | Day 1 compared to the 0th day (initial value)
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | Day 3 compared to the 0th day (initial value)
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | Day 5 compared to the 0th day (initial value)
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the collateral edema | Day 3 compared to the 0th day (initial value)
  Edema will be clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues).
Assessment of the collateral edema | Day 5 compared to the 0th day (initial value)
  Edema will be clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues)
Assessment of the collateral edema | Day 7 compared to the 0th day (initial value)
  Edema will be clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues).
Assessment of the quality of life | Day 7 compared to the 0th day (initial value)
  The patient's quality of life will be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire.
Assessment of the quality of life | Day 90-93 compared to the 0th day (initial value)
  The patient's quality of life will be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire.
Assessment of the quality of life | Day 180-186 compared to the 0th day (initial value)
  The patient's quality of life will be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire.
Doppler flowmetry | Day 7 compared to the 0th day (initial value)
  Doppler flowmetry will be carried out using the LAKK-02 apparatus (LLC Scientific and Production Enterprise "LAZMA" Russia) Registration certificate of the Ministry of Health of the Russian Federation No.29/03020703/5555-03 dated 11.09.2003).
Doppler flowmetry | Day 30-31 compared to the 0th day (initial value)
  Doppler flowmetry will be carried out using the LAKK-02 apparatus (LLC Scientific and Production Enterprise "LAZMA" Russia) Registration certificate of the Ministry of Health of the Russian Federation No.29/03020703/5555-03 dated 11.09.2003).
Doppler flowmetry | Day 90-93 compared to the 0th day (initial value)
  Doppler flowmetry will be carried out using the LAKK-02 apparatus (LLC Scientific and Production Enterprise "LAZMA" Russia) Registration certificate of the Ministry of Health of the Russian Federation No.29/03020703/5555-03 dated 11.09.2003).
Doppler flowmetry | Day 180-186 compared to the 0th day (initial value)
  Doppler flowmetry will be carried out using the LAKK-02 apparatus (LLC Scientific and Production Enterprise "LAZMA" Russia) Registration certificate of the Ministry of Health of the Russian Federation No.29/03020703/5555-03 dated 11.09.2003).
Histomorphometric analysis | Day 90-93 compared to the 0th day (initial value)
  Simultaneously with installation of gingiva formers, a soft tissue fragment is taken using a mucotome in the area of the previously performed mucous membrane thickness increasing for subsequent histomorphometric analysis. In the study, we use both conventional light microscopy (microscopy in the light field) and polarizing microscopy - to estimate the content of collagen fibers in preparations stained with picrosirius red. During a morphometric study, we carry out a quantitative assessment of the characteristics of the epithelial layer, the basement membrane relative length (the ratio of the absolute length of the basement membrane to the length of the epithelial layer), the characteristics of the underlying connective tissue.
Soft tissue aesthetics | Day 180-186 compared to the 0th day (initial value)
  Evaluation of soft tissue aesthetics will be carried out by visual inspection taking into account the PES (pink aesthetic score).
Keratinized mucosa width | Day 180-186 compared to the 0th day (initial value)
  Evaluation of the keratinized mucosa width will be carried out using a periodontal probe.
Probing depth | Day 180-186 compared to the 0th day (initial value)
  The probing depth will be carried out using a periodontal probe in the medial and distal papillae

CONTACTS AND LOCATIONS:
Overall Officials: Igor Ashurko, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
IPD Sharing is impossible because of the recommendation of the local ethics committee, the provision of data is possible upon receipt of an official request addressed to the chief researcher.